CLINICAL TRIAL: NCT01151657
Title: Probiotics for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Mejeribrugets ForskningsFond (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Luise Molenberg Begtrup, Doctor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MFF080409-2
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2009-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Irritable bowel syndrome; Probiotics; Treatment; Adequate relief
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Capsules containing maltodextrin.
  Interventions: Dietary Supplement: Placebo
- Probiotics (Experimental): Probiotics containing the 3 strains: Lactobacillus paracasei ssp paracasei F19, Lactobacillus acidophilus La5 og Bifidobacterium Bb12 in the dose of 2 x 109 - 10 x 109 CFU/capsule. The patients are to take 2x2 capsules a day.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Capsules with probiotics containing the strains : Lactobacillus paracasei ssp paracasei F19, Lactobacillus acidophilus La5 og Bifidobacterium Bb12. Dose/capsule : 2 x 109 - 10 x 109 CFU.
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo capsules containing maltodextrin
  Arms: Placebo

SUMMARY:
The study aims to investigate the effect of probiotics on IBS-patients symptoms compared to placebo, when given for 6 months.

By draw the investigators give IBS patients, in the age of 18-50 years, capsules with either probiotics or placebo. The patients are to take 2x2 capsules / day for 6 months. The patients are followed for 1 year. They are seen after 3, 6 and 12 months, and are followed by means of monthly letters.

The capsules contain 3 different probiotic strains - Lactobacillus paracasei ssp paracasei F19, Lactobacillus acidophilus La5 and Bifidobacterium Bb12. The dose is 2 x 109 - 10 x 109 CFU/capsule.

The hypothesis is, that there is a clinical difference between the group receiving probiotics and the group receiving placebo.

DETAILED DESCRIPTION:
Background: In management of IBS, no treatments have showed great efficacy. IBS is a non-fatal disease, so safety is a high priority in the choice of treatment. Probiotics is a dietary supplement and have no adverse effects. In some studies it has shown beneficial effect on some of the IBS patients symptoms, but some of the results are questionable. The studies have to be of longer duration, with more patients and the probiotics have to be capsules instead of milk based drinks.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ROME III criteria
* age 18-50 years
* signed informed content

Exclusion Criteria:

* Danger signals (fever, anaemia, weightloss, blod in stools, predisposition for CRC or IBD)
* abnormal physical examination
* comorbidity
* abuse
* lacking ability to talk and understand danish
* pregnancy
* For patients > 40 years. Changed bowel habits, with duration > 3 weeks, but < 1 year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Adequate relief | Every month for 12 months
  The patients are asked "In the last seven days, have you had adequate relief of your IBS symptoms?" . They are asked this question every month ( in a monthly letter) for 12 months.

SECONDARY OUTCOMES:
gastrointestinal symptoms | Every month for 12 months
  We use the questionnaires GSRS-IBS and GSRS. The patients are asked every month (in monthly letters) for 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ove B Schaffalitzky de Muckadell, Dr.Med, Professor, Principal Investigator — Department of gastroenterology, Odense University hospital
Locations (1):
- Research Unit for General Practice, Department of gastroenterology, Odense University hospital, Odense, Odense, Denmark

REFERENCES:
- [Derived] Begtrup LM, de Muckadell OB, Kjeldsen J, Christensen RD, Jarbol DE. Long-term treatment with probiotics in primary care patients with irritable bowel syndrome--a randomised, double-blind, placebo controlled trial. Scand J Gastroenterol. 2013 Oct;48(10):1127-35. doi: 10.3109/00365521.2013.825314. Epub 2013 Aug 19. PMID 23957590